CLINICAL TRIAL: NCT03506568
Title: A Universal Eye Drop Adherence Monitor to Measure and Improve Adherence to Ocular Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universal Adherence LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Oregon State University (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UniversalAdherence; 1R41EY028807-01 (NIH)
Record Dates: First submitted 2018-04-14; First posted 2018-04-24 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Medication Adherence; Glaucoma
Keywords: Adherence; Medication; Glaucoma; Device
MeSH Terms: conditions — Medication Adherence; Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control - no reminder (No Intervention): For Group 1, there will be no changes to their instructions or smart phone, which is the most common clinical situation.
- Integrated daily reminder using the D3 app (Experimental): For Group 2, they will have their D3 app turned on to deliver both a push notification reminder to their smart phone and audio and visual reminders to their D3 device.
  Interventions: Device: Devers Drop Device (D3) app

INTERVENTIONS:
Device: Devers Drop Device (D3) app — A universal eye drop cap monitor that accurately measures and improves eye drop-taking behavior.
  Arms: Integrated daily reminder using the D3 app

SUMMARY:
Glaucoma is the second leading cause of visual impairment worldwide. Eye drop medications reduce vision loss from glaucoma by at least 60%, but eye drops must be taken every day to be effective. However, adherence to eye drop treatment is poor with only 50% of patients regularly taking their prescribed eye drops. The investigators are developing the Devers Drop Device (D3) eye drop monitor to accurately measure eye drop cap removal and to improve eye drop-taking behavior. The investigators will test eye drop adherence with the D3 device in a randomized, prospective clinical trial.

DETAILED DESCRIPTION:
Universal Adherence is an emerging medical device company dedicated to improving adherence to ocular medications through innovative technical solutions. The Devers Drop Device (D3) will accurately track when a patient removes an eye drop bottle cap, communicate usage data wirelessly to a database that researchers can access, and send alerts to patients when a medication is due. In addition to helping patients maintain their dosing schedule, the D3 will also provide adherence information to researchers and eye care providers, which will help to understand poor treatment outcomes and to develop improved treatment strategies.The clinical benefits of the device in improving adherence will initially be assessed and targeted towards glaucoma, but the ability of the device to be attached to all FDA-approved eye drop bottle caps will make this device attractive to all patients that need consistent daily use of eye drops.

Randomized, prospective clinical trial: The investigators will enroll 50 participants (25 male, 25 female) into a prospective trial with duration of up to 50 days. The inclusion criteria are those who are prescribed latanoprost eye drop to be used once per day at bedtime, and own a functioning Android or Apple iphone smartphone (iOs) with Bluetooth and cellular connectivity. The investigators will exclude patients who currently use smartphone medication reminders and those with severe cognitive impairment limiting their ability to understand a questionnaire. The 50-day period is useful for glaucoma studies because patients revert to their normal dosing pattern within two weeks after their last visit. This study will include two stages: Stage 1) a 25-day period evaluating baseline patient adherence with the D3 device; and Stage 2) a subsequent 25-day period to determine the effect of no reminder versus daily reminder using the D3 app, which includes integrated audio and visual reminders.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are prescribed latanoprost eye drop to be used once per day at bedtime, and own a functioning smartphone and have a password-protected home wireless connection.

Exclusion Criteria:

* Patients who currently use smartphone medication reminders and those with severe cognitive impairment limiting their ability to understand a questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve L Mansberger, MD, Principal Investigator — Universal Adherence LLC; David Porter, PhD, Principal Investigator — Oregon State University
Locations (1):
- Robert Kinast, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared internally with co-investigators and those performing analysis of data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Baseline Adherence Test: During the initial testing to determine baseline adherence to the subject's glaucoma medication. If the subject's did not take their medication at least 90% of the time, they qualified to be randomized into the other 2 groups/arms
Period: Stage 1
Arm/Group | Control - no Reminder | Integrated Daily Reminder Using the D3 App | Baseline Adherence Test
Started | 0 | 0 | 50
Completed | 0 | 0 | 5
Not Completed | 0 | 0 | 45
Period: Stage 2
Arm/Group | Control - no Reminder | Integrated Daily Reminder Using the D3 App | Baseline Adherence Test
Started | 2 | 3 | 0
Completed | 1 | 2 | 0
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Adherence: Before randomizing subjects, all were given the device to observe if their adherence to their own medication was worse than 90% of the time. If so, they would enter the second stage and be placed in Group 1 or 2
- Total: Total of all reporting groups
Arm/Group | Control - no Reminder | Integrated Daily Reminder Using the D3 App | Baseline Adherence | Total
Number analyzed (Participants) | 2 | 3 | 45 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 12 | 14
  >=65 years | 2 | 1 | 33 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (6.36) | 64 (8.88) | 68.13 (11.17) | 67.8 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 18 | 21
  Male | 1 | 1 | 27 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 0 | 2 | 35 | 37
  African American | 1 | 1 | 1 | 3
  Hispanic | 1 | 0 | 1 | 2
  Asian or Pacific Islander | 0 | 0 | 8 | 8
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 45 | 50

OUTCOME MEASURES:

1. Primary Outcome: Compliance Percentage
Description: Compliance percentage by dividing the number of days the dose monitor recorded dosing within 3 hours of the prescribed time by the number of days in the study cycle
Time Frame: 50 days
Measure: Mean (Standard Deviation); unit: percentage of days dose monitor recorded
Groups:
- Baseline Adherence: All subjects received the device with no reminders and were monitored on how often they took their drops. If the drops were taken less than 90% of the required days, they were randomized to group 1 or 2
Arm/Group | Control - no Reminder | Integrated Daily Reminder Using the D3 App | Baseline Adherence
Number analyzed (Participants) | 1 | 2 | 50
percentage of days dose monitor recorded | 73.9 (NA) — Mean and Standard Deviation not available since only 1 participant was analyzed for the assessment | 94.6 (7.6) | 93.99 (16.2)

2. Secondary Outcome: Patient Satisfaction
Description: The investigators will also measure the participants' satisfaction with the dose monitor using a short Likert questionnaire. The questionnaire will include 5 questions. Each question will offer choices 1-5 with an overall minimum summed score of 5 and a maximum summed score of 25. Higher score will indicate higher satisfaction.
Time Frame: 50 days
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Baseline Adherence: Anyone who was not randomized into group 1 or 2 after taking their drops at least 90% of the time
Arm/Group | Control - no Reminder | Integrated Daily Reminder Using the D3 App | Baseline Adherence
Number analyzed (Participants) | 1 | 2 | 47
scores on a scale | 17 (NA) — Standard Deviation not available since only 1 participant was analyzed for the assessment | 22.5 (2.1) | 22.1 (3.0)

ADVERSE EVENTS:
Time Frame: 1 month
Description: The device does not change the level of risk for someone already taking eye drops.
Groups:
- Baseline Adherence: All subjects pre-randomization had the device with no reminders. If they took their eye drops at least 90% of the prescribed number of days they left the study
Arm/Group | Control - no Reminder | Integrated Daily Reminder Using the D3 App | Baseline Adherence
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 1/50
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/50
Other Adverse Events (participants affected / at risk) | 1/2 | 0/3 | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control - no Reminder (N=2) | Integrated Daily Reminder Using the D3 App (N=3) | Baseline Adherence (N=50)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Happened sometime during the month long period. Went away before returning to clinic. Believed to be non-serious and unrelated
Adenoviral Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Subject developed conjunctivitis unrelated to the study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT03506568/Prot_SAP_004.pdf
  • Informed Consent Form (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT03506568/ICF_003.pdf